CLINICAL TRIAL: NCT04206293
Title: Prospective, Open-Label Study, to Evaluate The Impact on Skin Quality Attributes by Juvederm® Volite Injection on Healthy Volunteers
Brief Title: A Study to Evaluate The Impact on Skin Quality Attributes by Juvederm® Volite Injection on Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CMO-MA-FAS-0617
Record Dates: First submitted 2019-12-18; First posted 2019-12-20 (Actual); Results first posted 2021-08-26 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-07

CONDITIONS: Healthy Adults; Skin Enhancement

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Juvéderm® VOLITE (Experimental): Participants received Juvéderm® VOLITE, intradermal injection on a zone of 8 centimeter (cm) x 4 cm (32 cm^2) of the volar left forearm on Day 0. The dose to be injected was decided by the investigator as per the Directions for Use. A maximum of 1 milliliter (mL) was injected on the zone treated.
  Interventions: Device: Juvederm® VOLITE

INTERVENTIONS:
Device: Juvederm® VOLITE — 1 mL of Juvéderm® VOLITE contains hyaluronic acid gel 12.0 milligram (mg), lidocaine hydrochloride 3.0 mg in a phosphate buffer pH 7.2 q.s. 1 mL (or gram).

SUMMARY:
To evaluate the impact on skin quality attributes, including physical measurements and gene and protein expression (histological and genomic analysis), following administration of Juvéderm® VOLITE in the volar forearms of healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants
* Participants with Fitzpatrick skin type II or III
* Participant willing to receive Juvéderm® VOLITE in the forearms and agrees to complete all study required procedures, including having 6 cutaneous punch biopsies taken in the forearms and blood drawn (Human immunodeficiency virus [HIV], B and C hepatitis analysis at screening)
* Written informed consent and data privacy consent obtained

Exclusion Criteria:

* Pregnant or nursing woman or planning a pregnancy during the study
* Participant participating to another research on human beings or being in an exclusion period for a previous study
* Intensive exposure to sunlight or ultraviolet (UV)-rays within the previous month and foreseen during the study
* Participant having other resorbable filling product injections, a laser treatment, an ultrasound-based treatment, radiation treatment, a dermabrasion, a surgery, a deep chemical peeling or other ablative procedure on the studied zones within the past 12 months prior to study start
* Participant with subcutaneous retaining structure on the studied zones (meshing, threads, gold strand)
* Participant having received injections of permanent or semi-permanent filling products in the studied zones
* Participant under anti-coagulant treatment or treatment liable to interfere with the healing process or hemostasis, during the previous month and during the study
* Participant receiving or is planning to receive anti-inflammatory drugs (oral/injectable corticosteroids or Nonsteroidal anti-inflammatory drugs (NSAIDs), e.g., aspirin, ibuprofen), or other substances known to increase coagulation time (herbal supplements with garlic or ginkgo biloba, etc) for 10 days prior to study treatment and 3 days after
* Participant under immunosuppressive therapy

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2020-07-29 (Actual); Study Completion 2020-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charlie Hee, Study Director — Allergan
Locations (1):
- EuroFins Dermscan Poland, Gdansk, Poland

RESULTS

PARTICIPANT FLOW:
Groups:
- Juvéderm® VOLITE Treated Zone: Participants received Juvéderm® VOLITE, intradermal injection on a zone of 8 cm x 4 cm (32 cm^2) of the volar left forearm on Day 0. The dose to be injected was decided by the investigator as per the Directions for Use. A maximum of 1 mL was injected on the zone treated.
Period: Overall Study
Arm/Group | Juvéderm® VOLITE Treated Zone
Started | 11
Completed | 10
Not Completed | 1
Not completed — Consent withdrawal | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set included any participant included in the study with at least a post-baseline value.
Arm/Group | Juvéderm® VOLITE Treated Zone
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.82 (6.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Skin Hydration (MoistureMeterD® XS Probe) [Mean (Standard Deviation); unit: tissue dielectric constant] — Skin hydration was measured using MoistureMeterD® XS (for epidermis and dermis), a non-invasive probe which measures the dielectric constant of the skin at a depth of 0.5 mm. 5 measurements were done on the same zone and the average value was calculated, expressed as tissue dielectric constant (TDC). The TDC is directly proportional to the amount of water in the tissue.
  tissue dielectric constant
    Juvéderm® VOLITE Treated Zone | 32.6 (4.3)
    Non-Treated Zone | 35.9 (5.3)
Skin Hydration (MoistureMeterD® S Probe) [Mean (Standard Deviation); unit: tissue dielectric constant] — Skin hydration was measured using MoistureMeter D® S15 (for epidermis and dermis), a non-invasive probe which measures the dielectric constant of the skin at a depth of 1.5 mm. 5 measurements were done on the same zone and the average value was calculated, expressed as TDC. The TDC is directly proportional to the amount of water in the tissue.
  tissue dielectric constant
    Juvéderm® VOLITE Treated Zone | 35.9 (5.3)
    Non-Treated Zone | 30.6 (2.6)
Skin Hydration (Corneometer®) [Mean (Standard Deviation); unit: arbitrary units of hydration] — Corneometer® measures the hydration level of the superficial skin surface (epidermis). It uses fringing field capacitance sensors to measure the dielectric constant of the skin. The dielectric constant of skin will change with water content. This allows for any changes in skin hydration to be measured by the precision measuring capacitor. These changes in water content of the stratum corneum are converted into arbitrary units of hydration. 5 measurements were done on the same zone and average value was calculated.
  arbitrary units of hydration
    Juvéderm® VOLITE Treated Zone | 29.5 (5.5)
    Non-Treated Zone | 29.3 (5.5)
Skin Elasticity Parameters (Cutometer ®) [Mean (Standard Deviation); unit: millimeters (mm)] — Skin elasticity was measured by a Cutometer ® which uses an in vivo non-invasive method to evaluate biological extensibility and elasticity variations. The various parameters analysed were Uf: final deformation (firmness), Ue: immediate extensibility, Ur: immediate retraction (tonicity), Ua: total recovery of the initial state. 2 measurements were done on the same zone and the average value was calculated.
  millimeters (mm)
    Uf: Juvéderm® VOLITE Treated Zone | 0.989 (0.109)
    Uf: Non-Treated Zone | 1.041 (0.127)
    Ue: Juvéderm® VOLITE Treated Zone | 0.816 (0.100)
    Ue: Non-Treated Zone | 0.864 (0.115)
    Ur: Juvéderm® VOLITE Treated Zone | 0.660 (0.131)
    Ur: Non-Treated Zone | 0.777 (0.138)
    Ua: Juvéderm® VOLITE Treated Zone | 0.844 (0.125)
    Ua: Non-Treated Zone | 0.916 (0.131)
Relative Parameters of Skin Elasticity (Cutometer ®) [Mean (Standard Deviation); unit: dimensionless] — The parameters evaluated were: Elastic Recovery (Q1)=elastic recovery area (QE)/maximum recovery area (QO), Viscous Recovery (Q2)=viscous recovery area (QR)/maximum recovery area (QO) and Viscoelastic Recovery (Q3)= (QE+QR)/QO. 2 measurements were done on the same zone and the average value was calculated.
  dimensionless
    Elastic Recovery (Q1): Juvéderm® VOLITE Treated Zone | 0.781 (0.052)
    Elastic Recovery (Q1): Non-Treated Zone | 0.825 (0.046)
    Viscous Recovery (Q2): Juvéderm® VOLITE Treated Zone | 0.630 (0.083)
    Viscous Recovery (Q2): Non-Treated Zone | 0.716 (0.073)
    Viscoelastic Recovery (Q3): Juvéderm® VOLITE Treated Zone | 0.151 (0.034)
    Viscoelastic Recovery (Q3): Non-Treated Zone | 0.109 (0.028)
Skin Elasticity [Mean (Standard Deviation); unit: Newton/meter] — Instant skin elasticity was measured with Elastimeter® and defines the skin elasticity determined as a resistance against deformation caused by the Elastimeter® probe on the skin surface. 3 measurements were done on the same zone and the average value was calculated. The values were expressed in Newton/meter.
  Newton/meter
    Juvéderm® VOLITE Treated Zone | 40.91 (10.27)
    Non-Treated Zone | 38.55 (11.49)
Skin Thickness (Skin Scanner®) [Mean (Standard Deviation); unit: mm] — Skin thickness was measured as the average thickness of the epidermis and dermis (in mm) using SkinScanner®, a high frequency echograph.
  mm
    Juvéderm® VOLITE Treated Zone | 1246 (160)
    Non-Treated Zone | 1064 (121)
Skin Density (Skin Scanner®) [Mean (Standard Deviation); unit: percentage of echogenic surface] — Skin density was measured as the percentage of echogenic surface using SkinScanner®, a high frequency echograph.
  percentage of echogenic surface
    Juvéderm® VOLITE Treated Zone | 33.63 (5.29)
    Non-Treated Zone | 44.05 (7.05)
Skin Roughness (Vivosight OCT®) [Mean (Standard Deviation); unit: micrometer (µm)] — Skin roughness was measured by Vivosight optical coherence tomography (OCT®) system which is used to obtain high resolution imaging of skin sub-structures and vascular networks. The skin roughness parameters from the images included Ra and Rz. Ra is a measure of the average length that is between peaks and valleys. Rz helps measure the vertical distance between the highest peak and the lowest valley.
  micrometer (µm)
    Ra: Juvéderm® VOLITE Treated Zone | 13.81 (2.99)
    Ra: Non-Treated Zone | 18.17 (2.16)
    Rz: Juvéderm® VOLITE Treated Zone | 89.50 (16.63)
    Rz: Non-Treated Zone | 111.73 (10.63)
Epidermal Thickness (Vivosight OCT®) [Mean (Standard Deviation); unit: µm] — Epidermal thickness is a skin density parameter measured by Vivosight OCT® system used to obtain high resolution imaging of skin sub-structures and vascular networks.
  µm
    Juvéderm® VOLITE Treated Zone | 92.64 (14.93)
    Non-Treated Zone | 94.58 (8.70)
Optical Attenuation Coefficient (OAC) (Vivosight OCT®) [Mean (Standard Deviation); unit: per mm (mm^-1)] — OAC is a skin density parameter measured by Vivosight OCT® system used to obtain high resolution imaging of skin sub-structures and vascular networks. It analytically describes the reduction of OCT signal intensity with increasing depth-in-tissue.
  per mm (mm^-1)
    Juvéderm® VOLITE Treated Zone | 2.61 (0.27)
    Non-Treated Zone | 2.71 (0.21)
Plexus Depth (Vivosight OCT®) [Mean (Standard Deviation); unit: µm] — Plexus depth is a skin vascularity parameter and was measured by Vivosight OCT® system which is used to obtain high resolution imaging of skin sub-structures and vascular networks.
  µm
    Juvéderm® VOLITE Treated Zone | 332.59 (13.90)
    Non-Treated Zone | 319.67 (17.84)
Vessel Diameter (Vivosight OCT®) [Mean (Standard Deviation); unit: µm] — Vessel diameter is a skin vascularity parameter and was measured by Vivosight OCT® system which is used to obtain high resolution imaging of skin sub-structures and vascular networks.
  µm
    Juvéderm® VOLITE Treated Zone | 44.13 (8.12)
    Non-Treated Zone | 46.64 (8.60)
Vessel Density [Mean (Standard Deviation); unit: dimensionless] — Vessel density is a skin vascularity parameter and was measured by Vivosight OCT® system which is used to obtain high resolution imaging of skin sub-structures and vascular networks.
  dimensionless
    Juvéderm® VOLITE Treated Zone | 1.98 (0.98)
    Non-Treated Zone | 2.24 (1.05)
300 μm Density [Mean (Standard Deviation); unit: dimensionless] — 300 μm density is a skin vascularity parameter and was measured by Vivosight OCT® system which is used to obtain high resolution imaging of skin sub-structures and vascular networks.
  dimensionless
    Juvéderm® VOLITE Treated Zone | 2.61 (0.62)
    Non-Treated Zone | 2.84 (0.70)
Skin Brightness Index [Mean (Standard Deviation); unit: glossymeter units] — Skin brightness index was measured using Glossymeter®. 3 measurements were done on the same zone and the average value was calculated. Values were expressed in "Glossymeter Units".
  glossymeter units
    Juvéderm® VOLITE Treated Zone | 6.3 (1.1)
    Non-Treated Zone | 5.7 (0.8)
Skin Colour (Spectrophotometer®) [Mean (Standard Deviation); unit: arbitrary units] — Skin colour was measured by Spectrophotometer®. It converts colours perceived by man to a digital code composed of three parameters: L*: for clarity (from dark to light) a*: for the green-to-red spectrum b*: for the blue-to-yellow spectrum; a* and b* are chrominance parameters, L* is a luminance parameter.
  arbitrary units
    a*: Juvéderm® VOLITE Treated Zone | 6.3 (2.0)
    a*: Non-Treated Zone | 7.0 (1.5)
    b*: Juvéderm® VOLITE Treated Zone | 17.2 (2.7)
    b*: Non-Treated Zone | 17.8 (2.3)
    L*: Juvéderm® VOLITE Treated Zone | 64.7 (2.8)
    L*: Non-Treated Zone | 64.1 (2.5)
Individual Typological Angle (ITA°) (Spectrophotometer®) [Mean (Standard Deviation); unit: degree] — Individual typological angle (ITA°), defines the skin pigmentation degree of a participant with taking into account the skin clarity (L*) and the melanin parameter (b*). 3 measurements were done on the same zone and the average values were calculated. Values are expressed in degree (°).
  degree
    Juvéderm® VOLITE Treated Zone | 40.5 (9.3)
    Non-Treated Zone | 38.4 (8.1)
Skin Melanin Index (Mexameter®) [Mean (Standard Deviation); unit: arbitrary units] — Melanin index measured with Mexameter® defines the skin pigmentation related to melanin content in the skin. Measurements are performed by the application of a probe to the skin surface. The probe has a 5 mm aperture that emits radiations. These radiations are reflected by the skin and captured back by the same probe. The results are expressed as an index value in arbitrary units from 0 to 999. 3 measurements were done on the same zone and the average value was calculated.
  arbitrary units
    Juvéderm® VOLITE Treated Zone | 150.03 (38.45)
    Non-Treated Zone | 181.40 (32.49)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Skin Hydration as Measured by MoistureMeterD® 0.5 mm
Description: Skin hydration was measured using MoistureMeterD® XS (for epidermis and dermis), a non-invasive probe which measures the dielectric constant of the skin at a depth of 0.5 mm. 5 measurements were done on the same zone and the average value was calculated, expressed as tissue dielectric constant (TDC). The TDC is directly proportional to the amount of water in the tissue. A positive change from Baseline indicates better skin hydration. Values were obtained from a mixed analysis of variance (ANOVA) model. The data is presented for area treated with Juvéderm® VOLITE and non-treated area in the same participants.
Time Frame: Baseline [Day 0 (D0)] to Days 28 (D28) and 84 (D84)
Population: Full Analysis Set (FAS) included any participant included in the study with at least a post-baseline value. Number analyzed is the number of participants with data available for analyses at the given timepoint.
Measure: Least Squares Mean (Standard Error); unit: tissue dielectric constant
Groups:
- Non-Treated Zone: The not-treated zone of the same arm in same the participant served as a control.
Arm/Group | Juvéderm® VOLITE Treated Zone | Non-Treated Zone
Number analyzed (Participants) | 11 | 11
tissue dielectric constant
  Change from Baseline to Day 28 | 1.7 (0.8) | -0.0 (0.7)
  Change from Baseline to Day 84: number analyzed (Participants) | 10 | 10
  Change from Baseline to Day 84 | 1.2 (0.9) | 0.6 (0.8)
Statistical Analysis 1: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Change from Baseline to Day 28; Test type: Superiority; p = 0.0736, Mixed ANOVA; Mixed ANOVA model was used for repeated measures with factors: Zone as fixed(treated,control),time as fixed(D0,D28,D84),zone by time interaction; Least Squares (LS) Mean Difference = 1.7, 95% CI 2-sided [-0.2 to 3.6], Standard Error of Mean 0.9
Statistical Analysis 2: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Change from Baseline to Day 84; Test type: Superiority; p = 0.5259, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 0.7, 95% CI 2-sided [-1.5 to 2.8], Standard Error of Mean 1.0

2. Primary Outcome: Change From Baseline in Skin Hydration as Measured by MoistureMeter D® 1.5 mm
Description: Skin hydration was measured using MoistureMeter D® S15 (for epidermis and dermis), a non-invasive probe which measures the dielectric constant of the skin at a depth of 1.5 mm. 5 measurements were done on the same zone and the average value was calculated, expressed as TDC. The TDC is directly proportional to the amount of water in the tissue. A positive change from Baseline indicates better skin hydration. Values were obtained from a mixed ANOVA model. The data is presented for area treated with Juvéderm® VOLITE and non-treated area in the same participants.
Time Frame: Baseline (D0) to D28 and D84
Population: FAS included any participant included in the study with at least a post-baseline value. Number analyzed is the number of participants with data available for analyses at the given timepoint.
Measure: Least Squares Mean (Standard Error); unit: tissue dielectric constant
Arm/Group | Juvéderm® VOLITE Treated Zone | Non-Treated Zone
Number analyzed (Participants) | 11 | 11
tissue dielectric constant
  Change from Baseline to Day 28 | 0.8 (1.3) | 1.0 (1.0)
  Change from Baseline to Day 84: number analyzed (Participants) | 10 | 10
  Change from Baseline to Day 84 | 1.4 (0.9) | 1.4 (0.6)
Statistical Analysis 1: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Change from Baseline to Day 28; Test type: Superiority; p = 0.8848, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.2, 95% CI 2-sided [-2.8 to 2.4], Standard Error of Mean 1.2
Statistical Analysis 2: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Change from Baseline to Day 84; Test type: Superiority; p = 0.9505, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-1.8 to 1.7], Standard Error of Mean 0.8

3. Primary Outcome: Change From Baseline in Skin Hydration as Measured by Corneometer®
Description: Corneometer® measures the hydration level of the superficial skin surface (epidermis). The measurement is based on capacitance measurement of a dielectric medium in this case skin. It uses fringing field capacitance sensors to measure the dielectric constant of the skin. The dielectric constant of skin will change with water content. This allows for any changes in skin hydration to be measured by the precision measuring capacitor. These changes in water content of the stratum corneum are converted into arbitrary units of hydration. 5 measurements were done on the same zone and average value was calculated. Values were obtained from a mixed ANOVA model and expressed in arbitrary units. A positive change from Baseline indicates better skin hydration rate. The data is presented for area treated with Juvéderm® VOLITE and non-treated area in the same participants.
Time Frame: Baseline (D0) to D28 and D84
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: arbitrary units of hydration
Arm/Group | Juvéderm® VOLITE Treated Zone | Non-Treated Zone
Number analyzed (Participants) | 11 | 11
arbitrary units of hydration
  Change from Baseline to Day 28 | 1.3 (1.1) | -1.4 (1.0)
  Change from Baseline to Day 84: number analyzed (Participants) | 10 | 10
  Change from Baseline to Day 84 | 2.5 (1.2) | 0.1 (1.2)
Statistical Analysis 1: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Change from Baseline to Day 28; Test type: Superiority; p = 0.0007, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 2.7, 95% CI 2-sided [1.4 to 4.0], Standard Error of Mean 0.6
Statistical Analysis 2: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Change from Baseline to Day 84; Test type: Superiority; p = 0.0033, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 2.4, 95% CI 2-sided [0.9 to 3.9], Standard Error of Mean 0.7

4. Primary Outcome: Change From Baseline in Skin Elasticity Parameters: Uf: Final Deformation (Firmness), Ue: Immediate Extensibility, Ur: Immediate Retraction (Tonicity), Ua: Total Recovery of the Initial State as Measured by Cutometer ®
Description: Skin elasticity was measured by a Cutometer ® which uses an in vivo non-invasive method to evaluate biological extensibility and elasticity variations. The various parameters analysed were Uf: final deformation (firmness), Ue: immediate extensibility, Ur: immediate retraction (tonicity), Ua: total recovery of the initial state. 2 measurements were done on the same zone and the average value was calculated. Values were obtained from a mixed ANOVA model. A Negative change from Baseline indicates firmer skin. The data is presented for area treated with Juvéderm® VOLITE and non-treated area in the same participants.
Time Frame: Baseline (D0) to D28 and D84
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Juvéderm® VOLITE Treated Zone | Non-Treated Zone
Number analyzed (Participants) | 11 | 11
mm
  Uf: Change from Baseline to Day 28 | -0.092 (0.009) | 0.003 (0.008)
  Uf: Change from Baseline to Day 84: number analyzed (Participants) | 10 | 10
  Uf: Change from Baseline to Day 84 | -0.073 (0.009) | -0.003 (0.007)
  Ue: Change from Baseline to Day 28 | -0.094 (0.010) | -0.005 (0.013)
  Ue: Change from Baseline to Day 84: number analyzed (Participants) | 10 | 10
  Ue: Change from Baseline to Day 84 | -0.075 (0.008) | 0.006 (0.009)
  Ur: Change from Baseline to Day 28 | -0.097 (0.015) | -0.018 (0.020)
  Ur: Change from Baseline to Day 84: number analyzed (Participants) | 10 | 10
  Ur: Change from Baseline to Day 84 | -0.096 (0.012) | -0.022 (0.015)
  Ua: Change from Baseline to Day 28 | -0.090 (0.015) | -0.009 (0.015)
  Ua: Change from Baseline to Day 84: number analyzed (Participants) | 10 | 10
  Ua: Change from Baseline to Day 84 | -0.093 (0.011) | -0.016 (0.010)
Statistical Analysis 1: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Uf: Change from Baseline to Day 28; Test type: Superiority; p < 0.0001, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.095, 95% CI 2-sided [-0.119 to -0.070], Standard Error of Mean 0.011
Statistical Analysis 2: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Uf: Change from Baseline to Day 84; Test type: Superiority; p < 0.0001, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.071, 95% CI 2-sided [-0.094 to -0.048], Standard Error of Mean 0.011
Statistical Analysis 3: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Ue: Change from Baseline to Day 28; Test type: Superiority; p < 0.0001, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.089, 95% CI 2-sided [-0.116 to -0.061], Standard Error of Mean 0.013
Statistical Analysis 4: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Ue: Change from Baseline to Day 84; Test type: Superiority; p < 0.0001, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.081, 95% CI 2-sided [-0.102 to -0.061], Standard Error of Mean 0.009
Statistical Analysis 5: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Ur: Change from Baseline to Day 28; Test type: Superiority; p = 0.0003, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.079, 95% CI [-0.116 to -0.041], Standard Error of Mean 0.018
Statistical Analysis 6: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Ur: Change from Baseline to Day 84; Test type: Superiority; p = 0.0001, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.074, 95% CI 2-sided [-0.103 to -0.044], Standard Error of Mean 0.013
Statistical Analysis 7: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Ua: Change from Baseline to Day 28; Test type: Superiority; p = 0.0002, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.081, 95% CI 2-sided [-0.117 to -0.045], Standard Error of Mean 0.017
Statistical Analysis 8: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Ua: Change from Baseline to Day 84; Test type: Superiority; p < 0.0001, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.077, 95% CI 2-sided [-0.103 to -0.052], Standard Error of Mean 0.012

5. Primary Outcome: Change From Baseline in Relative Parameters of Skin Elasticity: Q1, Q2, Q3 as Measured by Cutometer ®
Description: The parameters evaluated were: Elastic Recovery (Q1)=elastic recovery area (QE)/maximum recovery area (QO), Viscous Recovery (Q2)=viscous recovery area (QR)/maximum recovery area (QO) and Viscoelastic Recovery (Q3)= (QE+QR)/QO. 2 measurements were done on the same zone and the average value was calculated. Values were obtained from a mixed ANOVA model. A negative change from Baseline in Q1 and Q2 indicates decreased skin elasticity. A positive change from Baseline in Q3 indicates decreased skin elasticity. The data is presented for area treated with Juvéderm® VOLITE and non-treated area in the same participants.
Time Frame: Baseline (D0) to D28 and D84
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: dimensionless
Arm/Group | Juvéderm® VOLITE Treated Zone | Non-Treated Zone
Number analyzed (Participants) | 11 | 11
dimensionless
  Q1: Change from Baseline to Day 28 | -0.025 (0.015) | -0.017 (0.013)
  Q1: Change from Baseline to Day 84: number analyzed (Participants) | 10 | 10
  Q1: Change from Baseline to Day 84 | -0.042 (0.012) | -0.018 (0.011)
  Q2: Change from Baseline to Day 28 | -0.045 (0.017) | -0.023 (0.018)
  Q2: Change from Baseline to Day 84: number analyzed (Participants) | 10 | 10
  Q2: Change from Baseline to Day 84 | -0.053 (0.014) | -0.019 (0.015)
  Q3: Change from Baseline to Day 28 | 0.019 (0.006) | 0.006 (0.007)
  Q3: Change from Baseline to Day 84: number analyzed (Participants) | 10 | 10
  Q3: Change from Baseline to Day 84 | 0.013 (0.005) | 0.001 (0.006)
Statistical Analysis 1: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Q1: Change from Baseline to Day 28; Test type: Superiority; p = 0.5786, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.008, 95% CI 2-sided [-0.038 to 0.022], Standard Error of Mean 0.014
Statistical Analysis 2: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Q1: Change from Baseline to Day 84; Test type: Superiority; p = 0.0690, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.023, 95% CI 2-sided [-0.049 to 0.002], Standard Error of Mean 0.012
Statistical Analysis 3: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Q2: Change from Baseline to Day 28; Test type: Superiority; p = 0.1934, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.021, 95% CI 2-sided [-0.054 to 0.012], Standard Error of Mean 0.016
Statistical Analysis 4: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Q2: Change from Baseline to Day 84; Test type: Superiority; p = 0.0194, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.034, 95% CI 2-sided [-0.062 to -0.006], Standard Error of Mean 0.013
Statistical Analysis 5: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Q3: Change from Baseline to Day 28; Test type: Superiority; p = 0.0652, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 0.013, 95% CI 2-sided [-0.001 to 0.028], Standard Error of Mean 0.007
Statistical Analysis 6: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Q3: Change from Baseline to Day 84; Test type: Superiority; p = 0.0756, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 0.012, 95% CI 2-sided [-0.001 to 0.024], Standard Error of Mean 0.006

6. Secondary Outcome: Change From Baseline in Skin Elasticity as Measured by Elastimeter®
Description: Instant skin elasticity was measured with Elastimeter® and defines the skin elasticity determined as a resistance against deformation caused by the Elastimeter® probe on the skin surface. 3 measurements were done on the same zone and the average value was calculated. The values were expressed in Newton/meter. Higher values of ISE indicate higher skin elasticity. A positive change from Baseline indicates increased skin elasticity. Values were obtained from a mixed ANOVA model. The data is presented for area treated with Juvéderm® VOLITE and non-treated area in the same participants.
Time Frame: Baseline (D0) to D28 and D84
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Newton/meter
Arm/Group | Juvéderm® VOLITE Treated Zone | Non-Treated Zone
Number analyzed (Participants) | 11 | 11
Newton/meter
  Change from Baseline to Day 28 | 4.45 (2.12) | 5.00 (2.30)
  Change from Baseline to Day 84: number analyzed (Participants) | 10 | 10
  Change from Baseline to Day 84 | 3.90 (3.20) | 4.32 (3.49)
Statistical Analysis 1: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Change from Baseline to Day 28; Test type: Superiority; p = 0.8409, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.55, 95% CI 2-sided [-6.19 to 5.10], Standard Error of Mean 2.68
Statistical Analysis 2: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Change from Baseline to Day 84; Test type: Superiority; p = 0.9183, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.42, 95% CI 2-sided [-9.18 to 8.35], Standard Error of Mean 3.98

7. Secondary Outcome: Change From Baseline in Skin Thickness as Measured by Skin Scanner®
Description: Skin thickness was measured as the average thickness of the epidermis and dermis (in mm) using SkinScanner®, a high frequency echograph. Values were obtained from a mixed ANOVA model. A positive change from Baseline indicates increased skin thickness. The data is presented for area treated with Juvéderm® VOLITE and non-treated area in the same participants.
Time Frame: Baseline (D0) to D28 and D84
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Juvéderm® VOLITE Treated Zone | Non-Treated Zone
Number analyzed (Participants) | 11 | 11
mm
  Change from Baseline to Day 28 | 56 (72) | -14 (35)
  Change from Baseline to Day 84: number analyzed (Participants) | 10 | 10
  Change from Baseline to Day 84 | -85 (74) | -3 (36)
Statistical Analysis 1: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Change from Baseline to Day 28; Test type: Superiority; p = 0.4128, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 70, 95% CI 2-sided [-142 to 282], Standard Error of Mean 77
Statistical Analysis 2: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Change from Baseline to Day 84; Test type: Superiority; p = 0.3851, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -82, 95% CI 2-sided [-355 to 191], Standard Error of Mean 79

8. Secondary Outcome: Change From Baseline in Skin Density as Measured by Skin Scanner®
Description: Skin density was measured as the percentage of echogenic surface using SkinScanner®, a high frequency echograph. Values were obtained from a mixed ANOVA model. A positive change from Baseline indicates increased skin density. The data is presented for area treated with Juvéderm® VOLITE and non-treated area in the same participants.
Time Frame: Baseline (D0) to D28 and D84
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of echogenic surface
Arm/Group | Juvéderm® VOLITE Treated Zone | Non-Treated Zone
Number analyzed (Participants) | 11 | 11
percentage of echogenic surface
  Change from Baseline to Day 28 | 4.69 (2.82) | -1.83 (2.31)
  Change from Baseline to Day 84: number analyzed (Participants) | 10 | 10
  Change from Baseline to Day 84 | 8.56 (2.65) | 3.00 (2.27)
Statistical Analysis 1: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Change from Baseline to Day 28; Test type: Superiority; p = 0.0798, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 6.52, 95% CI 2-sided [-0.89 to 13.93], Standard Error of Mean 3.44
Statistical Analysis 2: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Change from Baseline to Day 84; Test type: Superiority; p = 0.1142, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 5.56, 95% CI 2-sided [-1.55 to 12.67], Standard Error of Mean 3.27

9. Secondary Outcome: Change From Baseline in Skin Roughness as Measured by Vivosight OCT®
Description: Skin roughness was measured by Vivosight optical coherence tomography (OCT®) system which is used to obtain high resolution imaging of skin sub-structures and vascular networks. The skin roughness parameters from the images included Ra and Rz. Ra is a measure of the average length that is between peaks and valleys. Rz helps measure the vertical distance between the highest peak and the lowest valley. Values were obtained from a mixed ANOVA model. A negative change from Baseline indicates decreased skin roughness. The data is presented for area treated with Juvéderm® VOLITE and non-treated area in the same participants.
Time Frame: Baseline (D0) to D28 and D84
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: µm
Arm/Group | Juvéderm® VOLITE Treated Zone | Non-Treated Zone
Number analyzed (Participants) | 11 | 11
µm
  Ra: Change from Baseline to Day 28 | -0.94 (0.64) | -1.90 (0.63)
  Ra: Change from Baseline to Day 84: number analyzed (Participants) | 10 | 10
  Ra: Change from Baseline to Day 84 | -0.27 (0.53) | -1.37 (0.54)
  Rz: Change from Baseline to Day 28 | -3.95 (3.59) | -9.85 (3.53)
  Rz: Change from Baseline to Day 84: number analyzed (Participants) | 10 | 10
  Rz: Change from Baseline to Day 84 | -3.64 (3.26) | -11.86 (3.35)
Statistical Analysis 1: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Ra: Change from Baseline to Day 28; Test type: Superiority; p = 0.2592, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 0.96, 95% CI 2-sided [-0.78 to 2.71], Standard Error of Mean 0.82
Statistical Analysis 2: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Ra: Change from Baseline to Day 84; Test type: Superiority; p = 0.1341, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 1.09, 95% CI 2-sided [-0.38 to 2.57], Standard Error of Mean 0.69
Statistical Analysis 3: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Rz: Change from Baseline to Day 28; Test type: Superiority; p = 0.2138, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 5.91, 95% CI 2-sided [-3.79 to 15.61], Standard Error of Mean 4.55
Statistical Analysis 4: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Rz: Change from Baseline to Day 84; Test type: Superiority; p = 0.0700, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 8.22, 95% CI 2-sided [-0.77 to 17.20], Standard Error of Mean 4.20

10. Secondary Outcome: Change From Baseline in Epidermal Thickness as Measured by Vivosight OCT®
Description: Epidermal thickness is a skin density parameter measured by Vivosight OCT® system used to obtain high resolution imaging of skin sub-structures and vascular networks. Values were obtained from a mixed ANOVA model. A positive change from Baseline indicates increased epidermal thickness. The data is presented for area treated with Juvéderm® VOLITE and non-treated area in the same participants.
Time Frame: Baseline (D0) to D28 and D84
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: µm
Arm/Group | Juvéderm® VOLITE Treated Zone | Non-Treated Zone
Number analyzed (Participants) | 11 | 11
µm
  Change from Baseline to Day 28 | 1.79 (2.80) | 1.68 (2.22)
  Change from Baseline to Day 84: number analyzed (Participants) | 10 | 10
  Change from Baseline to Day 84 | -1.93 (3.64) | -0.51 (2.77)
Statistical Analysis 1: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Change from Baseline to Day 28; Test type: Superiority; p = 0.9608, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 0.11, 95% CI 2-sided [-4.70 to 4.91], Standard Error of Mean 2.17
Statistical Analysis 2: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Change from Baseline to Day 84; Test type: Superiority; p = 0.6192, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -1.42, 95% CI 2-sided [-7.48 to 4.64], Standard Error of Mean 2.79

11. Secondary Outcome: Change From Baseline in Optical Attenuation Coefficient (OAC) as Measured by Vivosight OCT®
Description: OAC is a skin density parameter measured by Vivosight OCT® system used to obtain high resolution imaging of skin sub-structures and vascular networks. It analytically describes the reduction of OCT signal intensity with increasing depth-in-tissue. Values were obtained from a mixed ANOVA model. A positive change from Baseline indicates increased skin density. The data is presented for area treated with Juvéderm® VOLITE and non-treated area in the same participants.
Time Frame: Baseline (D0) to D28 and D84
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mm^-1
Arm/Group | Juvéderm® VOLITE Treated Zone | Non-Treated Zone
Number analyzed (Participants) | 11 | 11
mm^-1
  Change from Baseline to Day 28 | 0.02 (0.09) | 0.04 (0.08)
  Change from Baseline to Day 84: number analyzed (Participants) | 10 | 10
  Change from Baseline to Day 84 | 0.07 (0.07) | 0.18 (0.07)
Statistical Analysis 1: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Change from Baseline to Day 28; Test type: Superiority; p = 0.8322, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.02, 95% CI 2-sided [-0.20 to 0.16], Standard Error of Mean 0.08
Statistical Analysis 2: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Change from Baseline to Day 84; Test type: Superiority; p = 0.1334, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.11, 95% CI 2-sided [-0.25 to 0.04], Standard Error of Mean 0.07

12. Secondary Outcome: Change From Baseline in Plexus Depth as Measured by Vivosight OCT®
Description: Plexus depth is a skin vascularity parameter and was measured by Vivosight OCT® system which is used to obtain high resolution imaging of skin sub-structures and vascular networks. Values were obtained from a mixed ANOVA model. A negative change from Baseline indicates decreased plexus depth. The data is presented for area treated with Juvéderm® VOLITE and non-treated area in the same participants.
Time Frame: Baseline (D0) to D28 and D84
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: µm
Arm/Group | Juvéderm® VOLITE Treated Zone | Non-Treated Zone
Number analyzed (Participants) | 11 | 11
µm
  Change from Baseline to Day 28 | -11.54 (4.89) | -6.45 (6.52)
  Change from Baseline to Day 84: number analyzed (Participants) | 10 | 10
  Change from Baseline to Day 84 | -13.81 (5.07) | -20.55 (6.84)
Statistical Analysis 1: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Change from Baseline to Day 28; Test type: Superiority; p = 0.5221, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -5.09, 95% CI 2-sided [-21.56 to 11.38], Standard Error of Mean 7.78
Statistical Analysis 2: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Change from Baseline to Day 84; Test type: Superiority; p = 0.4174, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 6.74, 95% CI 2-sided [-10.55 to 24.03], Standard Error of Mean 8.07

13. Secondary Outcome: Change From Baseline in Vessel Diameter as Measured by Vivosight OCT®
Description: Vessel diameter is a skin vascularity parameter and was measured by Vivosight OCT® system which is used to obtain high resolution imaging of skin sub-structures and vascular networks. Values were obtained from a mixed ANOVA model. A positive change from Baseline indicates increased vessel diameter. The data is presented for area treated with Juvéderm® VOLITE and non-treated area in the same participants.
Time Frame: Baseline (D0) to D28 and D84
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: µm
Arm/Group | Juvéderm® VOLITE Treated Zone | Non-Treated Zone
Number analyzed (Participants) | 11 | 11
µm
  Change from Baseline to Day 28 | 2.59 (2.42) | -0.18 (2.62)
  Change from Baseline to Day 84: number analyzed (Participants) | 10 | 10
  Change from Baseline to Day 84 | 3.66 (2.35) | -6.33 (2.63)
Statistical Analysis 1: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Change from Baseline to Day 28; Test type: Superiority; p = 0.3052, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 2.77, 95% CI 2-sided [-2.90 to 8.44], Standard Error of Mean 2.58
Statistical Analysis 2: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Change from Baseline to Day 84; Test type: Superiority; p = 0.0016, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 9.99, 95% CI 2-sided [4.48 to 15.50], Standard Error of Mean 2.57

14. Secondary Outcome: Change From Baseline in Vessel Density as Measured by Vivosight OCT®
Description: Vessel density is a skin vascularity parameter and was measured by Vivosight OCT® system which is used to obtain high resolution imaging of skin sub-structures and vascular networks. A positive change from Baseline indicates increased vessel density. Values were obtained from a mixed ANOVA model. The data is presented for area treated with Juvéderm® VOLITE and non-treated area in the same participants.
Time Frame: Baseline (D0) to D28 and D84
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: dimensionless
Arm/Group | Juvéderm® VOLITE Treated Zone | Non-Treated Zone
Number analyzed (Participants) | 11 | 11
dimensionless
  Change from Baseline to Day 28 | 0.47 (0.50) | -0.23 (0.47)
  Change from Baseline to Day 84: number analyzed (Participants) | 10 | 10
  Change from Baseline to Day 84 | 0.19 (0.31) | -0.36 (0.30)
Statistical Analysis 1: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Change from Baseline to Day 28; Test type: Superiority; p = 0.1672, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 0.70, 95% CI 2-sided [-0.33 to 1.73], Standard Error of Mean 0.48
Statistical Analysis 2: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Change from Baseline to Day 84; Test type: Superiority; p = 0.0881, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 0.55, 95% CI 2-sided [-0.10 to 1.21], Standard Error of Mean 0.29

15. Secondary Outcome: Change From Baseline in 300 μm Density as Measured by Vivosight OCT®
Description: 300 μm density is a skin vascularity parameter and was measured by Vivosight OCT® system which is used to obtain high resolution imaging of skin sub-structures and vascular networks. Values were obtained from a mixed ANOVA model. A positive change from Baseline indicates increased 300 μm density. The data is presented for area treated with Juvéderm® VOLITE and non-treated area in the same participants.
Time Frame: Baseline (D0) to D28 and D84
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: dimensionless
Arm/Group | Juvéderm® VOLITE Treated Zone | Non-Treated Zone
Number analyzed (Participants) | 11 | 11
dimensionless
  Change from Baseline to Day 28 | 0.75 (0.26) | 0.17 (0.31)
  Change from Baseline to Day 84: number analyzed (Participants) | 10 | 10
  Change from Baseline to Day 84 | 0.13 (0.29) | 0.33 (0.34)
Statistical Analysis 1: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Change from Baseline to Day 28; Test type: Superiority; p = 0.0577, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 0.57, 95% CI 2-sided [-0.02 to 1.17], Standard Error of Mean 0.28
Statistical Analysis 2: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Change from Baseline to Day 84; Test type: Superiority; p = 0.5224, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.20, 95% CI 2-sided [-0.85 to 0.45], Standard Error of Mean 0.31

16. Secondary Outcome: Change From Baseline in Skin Brightness Index as Measured by Glossymeter®
Description: Skin brightness index was measured using Glossymeter®. 3 measurements were done on the same zone and the average value was calculated. Values were expressed in "Glossymeter Units". Values were obtained from a mixed ANOVA model. Higher glossymeter values indicate higher skin brightness. A positive change from Baseline indicates increased skin brightness. The data is presented for area treated with Juvéderm® VOLITE and non-treated area in the same participants.
Time Frame: Baseline (D0) to D28 and D84
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: glossymeter unit
Arm/Group | Juvéderm® VOLITE Treated Zone | Non-Treated Zone
Number analyzed (Participants) | 11 | 11
glossymeter unit
  Change from Baseline to Day 28 | 0.1 (0.2) | 0.3 (0.1)
  Change from Baseline to Day 84: number analyzed (Participants) | 10 | 10
  Change from Baseline to Day 84 | 0.4 (0.2) | 0.2 (0.2)
Statistical Analysis 1: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Change from Baseline to Day 28; Test type: Superiority; p = 0.2666, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.2, 95% CI 2-sided [-0.6 to 0.2], Standard Error of Mean 0.2
Statistical Analysis 2: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Change from Baseline to Day 84; Test type: Superiority; p = 0.4366, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 0.2, 95% CI 2-sided [-0.3 to 0.7], Standard Error of Mean 0.2

17. Secondary Outcome: Change From Baseline in Skin Colour as Measured by Spectrophotometer®
Description: Skin colour was measured by Spectrophotometer®. It converts colours perceived by man to a digital code composed of three parameters: L*: for clarity (from dark to light) a*: for the green-to-red spectrum b*: for the blue-to-yellow spectrum; a* and b* are chrominance parameters, L* is a luminance parameter. Higher values of a*, b*and L* indicates 'skin more red', 'skin more yellow' and 'skin clearer'. Values were obtained from a mixed ANOVA model and expressed in arbitrary units. The data is presented for area treated with Juvéderm® VOLITE and non-treated area in the same participants.
Time Frame: Baseline (D0) to D28 and D84
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: arbitrary units
Arm/Group | Juvéderm® VOLITE Treated Zone | Non-Treated Zone
Number analyzed (Participants) | 11 | 11
arbitrary units
  a*: Change from Baseline to Day 28 | -0.3 (0.2) | -0.1 (0.2)
  a*: Change from Baseline to Day 84: number analyzed (Participants) | 10 | 10
  a*: Change from Baseline to Day 84 | 0.8 (0.3) | -0.7 (0.2)
  b*: Change from Baseline to Day 28 | -0.3 (0.3) | -0.2 (0.2)
  b*: Change from Baseline to Day 84: number analyzed (Participants) | 10 | 10
  b*: Change from Baseline to Day 84 | -1.4 (0.4) | -1.1 (0.4)
  L*: Change from Baseline to Day 28 | 0.4 (0.3) | 0.8 (0.3)
  L*: Change from Baseline to Day 84: number analyzed (Participants) | 10 | 10
  L*: Change from Baseline to Day 84 | 0.7 (0.3) | 1.1 (0.3)
Statistical Analysis 1: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; a*: Change from Baseline to Day 28; Test type: Superiority; p = 0.4197, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.2, 95% CI 2-sided [-0.6 to 0.3], Standard Error of Mean 0.2
Statistical Analysis 2: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; a*: Change from Baseline to Day 84; Test type: Superiority; p = 0.9140, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.0, 95% CI 2-sided [-0.6 to 0.5], Standard Error of Mean 0.3
Statistical Analysis 3: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; b*: Change from Baseline to Day 28; Test type: Superiority; p = 0.7604, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.6 to 0.4], Standard Error of Mean 0.2
Statistical Analysis 4: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; b*: Change from Baseline to Day 84; Test type: Superiority; p = 0.5936, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.2, 95% CI 2-sided [-1.0 to 0.6], Standard Error of Mean 0.4
Statistical Analysis 5: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; L*: Change from Baseline to Day 28; Test type: Superiority; p = 0.0808, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.4, 95% CI 2-sided [-0.9 to 0.1], Standard Error of Mean 0.2
Statistical Analysis 6: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; L*: Change from Baseline to Day 84; Test type: Superiority; p = 0.1633, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.4, 95% CI 2-sided [-1.0 to 0.2], Standard Error of Mean 0.3

18. Secondary Outcome: Change From Baseline in Individual Typological Angle (ITA°) as Measured by Spectrophotometer®
Description: Individual typological angle (ITA°), defines the skin pigmentation degree of a participant with taking into account the skin clarity (L*) and the melanin parameter (b*). 3 measurements were done on the same zone and the average values were calculated. Values were obtained from a mixed ANOVA model and expressed in degree (°). Higher values of ITA° indicates 'skin less pigmented'. A positive change from Baseline indicates less pigmented skin. The data is presented for area treated with Juvéderm® VOLITE and non-treated area in the same participants.
Time Frame: Baseline (D0) to D28 and D84
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: degree
Arm/Group | Juvéderm® VOLITE Treated Zone | Non-Treated Zone
Number analyzed (Participants) | 11 | 11
degree
  Change from Baseline to Day 28 | 1.4 (0.6) | 2.0 (0.5)
  Change from Baseline to Day 84: number analyzed (Participants) | 10 | 10
  Change from Baseline to Day 84 | 3.8 (1.2) | 4.0 (1.0)
Statistical Analysis 1: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Change from Baseline to Day 28; Test type: Superiority; p = 0.1977, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.6, 95% CI 2-sided [-1.6 to 0.4], Standard Error of Mean 0.4
Statistical Analysis 2: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Change from Baseline to Day 84; Test type: Superiority; p = 0.7535, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.3, 95% CI 2-sided [-2.2 to 1.7], Standard Error of Mean 0.9

19. Secondary Outcome: Change From Baseline in Skin Melanin Index as Measured by Mexameter®
Description: Melanin index measured with Mexameter® defines the skin pigmentation related to melanin content in the skin. Measurements are performed by the application of a probe to the skin surface. The probe has a 5 mm aperture that emits radiations. These radiations are reflected by the skin and captured back by the same probe. The results are expressed as an index value for each parameter in arbitrary units from 0 to 999. 3 measurements were done on the same zone and the average value was calculated. Values were obtained from a mixed ANOVA model. A negative change from Baseline indicates less pigmented skin. The data is presented for area treated with Juvéderm® VOLITE and non-treated area in the same participants.
Time Frame: Baseline (D0) to D28 and D84
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: arbitrary units
Arm/Group | Juvéderm® VOLITE Treated Zone | Non-Treated Zone
Number analyzed (Participants) | 11 | 11
arbitrary units
  Change from Baseline to Day 28 | -3.78 (4.66) | -8.13 (3.34)
  Change from Baseline to Day 84: number analyzed (Participants) | 10 | 10
  Change from Baseline to Day 84 | -2.53 (7.44) | -19.79 (5.47)
Statistical Analysis 1: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Change from Baseline to Day 28; Test type: Superiority; p = 0.2905, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 4.35, 95% CI 2-sided [-4.16 to 12.85], Standard Error of Mean 3.95
Statistical Analysis 2: Comparison: Juvéderm® VOLITE Treated Zone vs Non-Treated Zone; Change from Baseline to Day 84; Test type: Superiority; p = 0.0241, Mixed ANOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 17.27, 95% CI 2-sided [2.84 to 31.69], Standard Error of Mean 6.37

20. Primary Outcome: Number of Participants With at Least One Treatment-emergent Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. A treatment-emergent AE is an AE that occurs or worsens after a participant receives study drug.
Time Frame: First dose of study treatment to end of the study (Up to 9 months)
Population: Safety Population included any participant having used the tested device.
Measure: Count of Participants; unit: Participants
Arm/Group | Juvéderm® VOLITE Treated Zone
Number analyzed (Participants) | 11
Participants | 5

21. Secondary Outcome: Number of Participants With Injection Site Reactions (ISR)
Description: ISRs are reactions that occur after injection of the study drug. The following ISRs: Redness/Erythema, Pain/Tenderness, Induration, Swelling/Oedema, Lumps/Bumps, Bruising/Hematoma, Itching, Discoloration/Pigmentation were reported as None, Mild, Moderate or Severe. Only those categories reported for at least 1 participant are reported.
Time Frame: Day 0
Population: Safety Population included any participant having used the tested device.
Measure: Count of Participants; unit: Participants
Arm/Group | Juvéderm® VOLITE Treated Zone
Number analyzed (Participants) | 11
Participants
  Redness/Erythema: Mild | 11
  Pain/Tenderness: None | 4
  Pain/Tenderness: Mild | 7
  Induration: None | 11
  Swelling/Oedema: None | 4
  Swelling/Oedema: Mild | 7
  Lumps/Bumps: None | 3
  Lumps/Bumps: Mild | 8
  Bruising/Hematoma: None | 4
  Bruising/Hematoma: Mild | 6
  Bruising/Hematoma: Moderate | 1
  Itching: None | 11
  Discoloration/Pigmentation: None | 11

ADVERSE EVENTS:
Time Frame: First dose of study treatment to end of the study (Up to 9 months)
Description: All-Cause Mortality included all randomized participants. Serious Adverse Events and Other Adverse Events: Safety Population included any participant having used the tested device.
Arm/Group | Juvéderm® VOLITE Treated Zone
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 5/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Juvéderm® VOLITE Treated Zone (N=11)
Diarrhea (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Oedema (General disorders) | 3
Pain (General disorders) | 2
Herpes virus infection (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 2
Burning sensation (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Skin tightness (Skin and subcutaneous tissue disorders) | 2
Haematoma (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2019-08-21): https://cdn.clinicaltrials.gov/large-docs/93/NCT04206293/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-16): https://cdn.clinicaltrials.gov/large-docs/93/NCT04206293/SAP_001.pdf